CLINICAL TRIAL: NCT02291029
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CFZ533 in Patients With Primary Sjögren's Syndrome
Brief Title: Safety, Pharmacokinetics and Preliminary Efficacy Study of CFZ533 in Patients With Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCFZ533X2203
Record Dates: First submitted 2014-11-04; First posted 2014-11-14 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-07

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Sjögren's syndrome, CFZ533, ESSDAI
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- CFZ533 active- Cohort 2 (Experimental): multiple doses of CFZ533 intravenous infusion
  Interventions: Drug: CFZ533 active - Cohort 2
- CFZ533 placebo- Cohort 2 (Placebo Comparator): multiple doses of placebo intravenous infusion
  Interventions: Drug: CFZ533 placebo - Cohort 2
- CFZ533 active - Cohort 1 (Experimental): multiple doses of CFZ533 s.c. injection
  Interventions: Drug: CFZ533 active - Cohort 1
- CFZ533 placebo - Cohort 1 (Placebo Comparator): multiple doses of placebo s.c. injection
  Interventions: Drug: CFZ533 placebo- Cohort 1
- CFZ533 Treatment Arm 1 - Cohort 3 (Experimental): multiple doses of CFZ533 s.c. injection
  Interventions: Drug: CFZ533 active -Cohort 3
- CFZ533 Treatment Arm 2 - Cohort 3 (Experimental): Single dose of CFZ533 i.v. infusion and multiple doses of CFZ533 s.c. injection
  Interventions: Drug: CFZ533 active - Cohort 3

INTERVENTIONS:
Drug: CFZ533 active - Cohort 1 — multiple doses of CFZ533 s.c. injection
  Arms: CFZ533 active - Cohort 1
Drug: CFZ533 placebo- Cohort 1 — multiple doses of placebo s.c. injection
  Arms: CFZ533 placebo - Cohort 1
Drug: CFZ533 active - Cohort 2 — multiple doses of CFZ533 intravenous infusion
  Arms: CFZ533 active- Cohort 2
Drug: CFZ533 placebo - Cohort 2 — multiple doses of placebo intravenous infusion
  Arms: CFZ533 placebo- Cohort 2
Drug: CFZ533 active -Cohort 3 — multiple doses of CFZ533 s.c. injection
  Arms: CFZ533 Treatment Arm 1 - Cohort 3
Drug: CFZ533 active - Cohort 3 — Single dose of CFZ533 i.v. infusion and multiple doses of CFZ533 s.c. injection
  Arms: CFZ533 Treatment Arm 2 - Cohort 3

SUMMARY:
This study did evaluate the safety,tolerability and preliminary therapeutic efficacy of multiple doses of intravenous infusion of CFZ533 monoclonal antibody in patients with primary Sjögren's syndrome(pSS)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Sjögren's syndrome
* ESSDAI score ≥ 6

Exclusion Criteria:

* Secondary Sjögren's syndrome
* Receiving cyclosphosphamide, corticosteroid bolus with dose over 1 mg/kg, rituximab, belimunab, other immunosuppressives.
* At significant risk for thromboembolic event
* Clinically significant systemic infection
* Significant elevated risk for infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (3):
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, Duncansville, Pennsylvania
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Debrecen, Hungary
- Novartis Investigative Site, Basel, Switzerland
- United Kingdom (3):
  - Novartis Investigative Site, Edgbaston, Birmingham
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Fisher BA, Szanto A, Ng WF, Bombardieri M, Posch MG, Papas AS, Farag AM, Daikeler T, Bannert B, Kyburz D, Kivitz AJ, Carsons SE, Isenberg DA, Barone F, Bowman SJ, Espie P, Floch D, Dupuy C, Ren X, Faerber PM, Wright AM, Hockey HU, Rotte M, Milojevic J, Avrameas A, Valentin MA, Rush JS, Gergely P. Assessment of the anti-CD40 antibody iscalimab in patients with primary Sjogren's syndrome: a multicentre, randomised, double-blind, placebo-controlled, proof-of-concept study. Lancet Rheumatol. 2020 Mar;2(3):e142-e152. doi: 10.1016/S2665-9913(19)30135-3. Epub 2020 Jan 23. PMID 38263652
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 69 patients were enrolled in Germany (1 center), Hungary (1 center), Switzerland (1 center), United Kingdom (3 centers), United States (3 centers)
Groups:
- Cohort 1 CFZ533: CFZ533 3 mg/kg s.c.
- Cohort 1 Placebo: Placebo s.c./CFZ533 3 mg/kg s.c.
- Cohort 2 CFZ533: CFZ533 10 mg/kg i.v.
- Cohort 2 Placebo: Placebo i.v./CFZ533 10 mg/kg i.v.
- Cohort 3 CFZ533 Arm 1: CFZ533 600 mg s.c./CFZ533 300 mg s.c.
- Cohort 3 CFZ533 Arm 2: CFZ533 10 mg/kg i.v./CFZ533 300 mg s.c.
Period: Overall Study
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo | Cohort 3 CFZ533 Arm 1 | Cohort 3 CFZ533 Arm 2
Started | 8 | 4 | 21 | 11 | 13 | 12
Completed | 8 | 3 | 20 | 11 | 13 | 12
Not Completed | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo | Cohort 3 CFZ533 Arm 1 | Cohort 3 CFZ533 Arm 2 | Total
Number analyzed (Participants) | 8 | 4 | 21 | 11 | 13 | 12 | 69
Age, Continuous [Mean (Full Range); unit: years] | 56.4 [34 to 72] | 48.8 [45 to 52] | 51.7 [24 to 72] | 50.6 [25 to 69] | 52.3 [23 to 74] | 54.8 [23 to 68] | 52.6 [23 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 19 | 11 | 12 | 10 | 64
  Male | 0 | 0 | 2 | 0 | 1 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7 | 4 | 18 | 10 | 12 | 10 | 61
  Asian | 1 | 0 | 2 | 1 | 1 | 2 | 7
  Black | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI)
Description: The effect of CFZ533 on clinical disease activity was measured by the change in ESSDAI (EULAR Sjögren's syndrome disease activity index) between baseline and week 12. The instrument contains 12 organ-specific domains contributing to disease activity. For each domain, features of disease activity are scored in 3 or 4 levels according to their severity.
  These scores are then summed across the 12 domains in a weighted manner to provide the total score (range 0-123). A reduction from baseline indicates improvement in patients.
Time Frame: Baseline and Week 12
Population: PD Population (all subjects with available Pharmacodynamics data and no protocol deviations with relevant impact on PD data)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo | Cohort 3 CFZ533 Arm 1 | Cohort 3 CFZ533 Arm 2
Number analyzed (Participants) | 8 | 4 | 21 | 11 | 13 | 12
units on a scale
  Baseline | 12.0 (3.78) | 11.8 (3.86) | 10.6 (4.44) | 11.0 (5.16) | 12.7 (6.06) | 10.4 (5.87)
  Week 12: number analyzed (Participants) | 8 | 4 | 20 | 11 | 13 | 12
  Week 12 | 9.6 (5.45) | 9.8 (3.30) | 4.2 (4.25) | 9.7 (9.05) | 7.2 (6.69) | 2.8 (2.48)
  Change from Baseline to Week 12: number analyzed (Participants) | 8 | 4 | 20 | 11 | 13 | 12
  Change from Baseline to Week 12 | -2.4 (2.77) | -2.0 (2.45) | -6.4 (4.00) | -1.3 (8.06) | -5.5 (5.49) | -7.6 (7.14)
Statistical Analysis 1: Comparison: Cohort 1 CFZ533 vs Cohort 1 Placebo; Test type: Superiority; p = 0.397, Repeated measures model — One-sided p-value; with time (as nominal study week), the interaction between time and treatment (all as fixed effects) and with baseline as a covariate; Mean Difference (Net) = -0.41, 95% CI 2-sided [-3.70 to 2.89]
Statistical Analysis 2: Comparison: Cohort 2 CFZ533 vs Cohort 2 Placebo; Test type: Superiority; p = 0.009, Repeated measures model — One-sided p-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -5.21, 95% CI 2-sided [-9.46 to -0.96]
Statistical Analysis 3: Comparison: Cohort 3 CFZ533 Arm 1 vs Cohort 3 CFZ533 Arm 2; Test type: Superiority; p = 0.344, Repeated measures model — two-sided p-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.34, 95% CI 2-sided [-2.78 to 7.45]

2. Secondary Outcome: Change From Baseline in EULAR Sjögren's Syndrome Patient Reported Intensity (ESSPRI)
Description: The ESSPRI is a patient self-reported outcome measure to assess dryness, limb pain, fatigue and mental fatigue, where each of the domains normally reported as 0 (not at all) to 10 (extremely severe). The final ESSPRI score is the average of three: dryness, pain and fatigue. A reduction from baseline indicates the improvement of symptoms.
Time Frame: Baseline and Week 12
Population: PD Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo | Cohort 3 CFZ533 Arm 1 | Cohort 3 CFZ533 Arm 2
Number analyzed (Participants) | 8 | 4 | 21 | 11 | 13 | 12
units on a scale
  Baseline | 6.75 (1.909) | 7.00 (1.826) | 6.71 (1.678) | 7.18 (1.486) | 7.00 (1.604) | 6.00 (2.344)
  Week 12: number analyzed (Participants) | 8 | 4 | 20 | 11 | 13 | 12
  Week 12 | 5.71 (1.240) | 7.08 (2.251) | 5.03 (2.413) | 6.24 (2.039) | 5.33 (2.269) | 4.83 (2.552)
  Change from Baseline to Week 12: number analyzed (Participants) | 8 | 4 | 20 | 11 | 13 | 12
  Change from Baseline to Week 12 | -1.04 (1.201) | 0.08 (0.631) | -1.68 (1.954) | -0.94 (1.246) | -1.67 (1.841) | -1.17 (2.333)
Statistical Analysis 1: Comparison: Cohort 1 CFZ533 vs Cohort 1 Placebo; Test type: Superiority; p = 0.205, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.09, 95% CI 2-sided [-2.97 to 0.80]
Statistical Analysis 2: Comparison: Cohort 2 CFZ533 vs Cohort 2 Placebo; Test type: Superiority; p = 0.188, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.95, 95% CI 2-sided [-2.41 to 0.50]
Statistical Analysis 3: Comparison: Cohort 3 CFZ533 Arm 1 vs Cohort 3 CFZ533 Arm 2; Test type: Superiority; p = 0.663, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.37, 95% CI 2-sided [-2.08 to 1.35]

3. Secondary Outcome: Change From Baseline in Physician Global Assessment of the Patient's Overall Disease Activity (VAS)
Description: The visual analogue scale used is a 100 mm VAS ranging from "no disease" (0 mm) to "maximal disease activity" (100 mm).
Time Frame: Baseline and Week 12
Population: PD Population (Statistical Analysis only for Cohort 1 and 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo | Cohort 3 CFZ533 Arm 1 | Cohort 3 CFZ533 Arm 2
Number analyzed (Participants) | 8 | 4 | 21 | 11 | 13 | 12
units on a scale
  Baseline: number analyzed (Participants) | 7 | 4 | 21 | 11 | 13 | 12
  Baseline | 57.9 (15.72) | 57.8 (17.19) | 51.9 (12.62) | 47.9 (19.18) | 50.4 (12.39) | 47.1 (18.34)
  Week 12: number analyzed (Participants) | 8 | 4 | 20 | 11 | 13 | 12
  Week 12 | 40.5 (16.42) | 55.5 (12.01) | 22.8 (11.78) | 34.2 (13.90) | 25.4 (16.65) | 27.3 (16.74)
  Change from Baseline to Week 12: number analyzed (Participants) | 7 | 4 | 20 | 11 | 13 | 12
  Change from Baseline to Week 12 | -17.6 (24.60) | -2.3 (10.90) | -28.7 (16.02) | -13.7 (22.97) | -25.0 (15.30) | -19.8 (21.96)
Statistical Analysis 1: Comparison: Cohort 1 CFZ533 vs Cohort 1 Placebo; Test type: Superiority; p = 0.161, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -15.26, 95% CI 2-sided [-37.90 to 7.38]
Statistical Analysis 2: Comparison: Cohort 2 CFZ533 vs Cohort 2 Placebo; Test type: Superiority; p = 0.017, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -12.16, 95% CI 2-sided [-21.94 to -2.38]

4. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Their Disease Activity (VAS)
Description: The visual analogue scale used is a 100 mm VAS ranging from "no disease" (0 mm) to "maximal disease activity" (100 mm).
Time Frame: Baseline and Week 12
Population: PD Population (Statistical Analysis only for Cohort 1 and 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo | Cohort 3 CFZ533 Arm 1 | Cohort 3 CFZ533 Arm 2
Number analyzed (Participants) | 8 | 4 | 21 | 11 | 13 | 12
units on a scale
  Baseline | 47.13 (32.406) | 73.00 (12.623) | 58.43 (19.881) | 54.91 (21.002) | 63.69 (25.799) | 52.08 (22.138)
  Week 12: number analyzed (Participants) | 8 | 4 | 20 | 11 | 13 | 12
  Week 12 | 49.06 (24.519) | 75.50 (24.393) | 34.85 (24.564) | 42.27 (24.483) | 38.46 (26.965) | 53.17 (25.305)
  Change from Baseline to Week 12: number analyzed (Participants) | 8 | 4 | 20 | 11 | 13 | 12
  Change from Baseline to Week 12 | 1.94 (26.023) | 2.50 (17.861) | -23.05 (26.920) | -12.64 (26.871) | -25.23 (29.833) | 1.08 (23.283)
Statistical Analysis 1: Comparison: Cohort 1 CFZ533 vs Cohort 1 Placebo; Test type: Superiority; p = 0.456, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -9.45, 95% CI 2-sided [-36.20 to 17.30]
Statistical Analysis 2: Comparison: Cohort 2 CFZ533 vs Cohort 2 Placebo; Test type: Superiority; p = 0.376, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -8.14, 95% CI 2-sided [-26.67 to 10.39]

5. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Physical Component Score
Description: The SF-36 is a 36-item, patient self-reported outcome measure (questionnaires) of patient health. The outcome of the questionnaires in eight scales results in two summary scores, physical component and mental component, both ranging from 0 - 100. An increase from baseline in either component summary score indicates reduced disease burden.
Time Frame: Baseline and Week 12
Population: PD Population for Cohort 1 and Cohort 2. Data were not collected from participants in Cohort 3 CFZ533 Arm 1 and Cohort 3 CFZ533 Arm 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo
Number analyzed (Participants) | 8 | 4 | 21 | 11
units on a scale
  Baseline: number analyzed (Participants) | 6 | 4 | 20 | 11
  Baseline | 42.218 (6.9437) | 31.215 (12.5562) | 38.163 (8.5905) | 38.819 (5.9689)
  Week 12: number analyzed (Participants) | 8 | 4 | 18 | 11
  Week 12 | 40.374 (9.2230) | 36.123 (13.0002) | 44.001 (9.3943) | 40.298 (8.9392)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 4 | 17 | 11
  Change from Baseline to Week 12 | -1.005 (4.5380) | 4.908 (4.2349) | 5.546 (7.1760) | 1.479 (8.2497)
Statistical Analysis 1: Comparison: Cohort 1 CFZ533 vs Cohort 1 Placebo; Test type: Superiority; p = 0.172, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -5.50, 95% CI 2-sided [-13.91 to 2.91]
Statistical Analysis 2: Comparison: Cohort 2 CFZ533 vs Cohort 2 Placebo; Test type: Superiority; p = 0.175, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 3.83, 95% CI 2-sided [-1.81 to 9.48]

6. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Mental Component Score
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo
Number analyzed (Participants) | 8 | 4 | 21 | 11
units on a scale
  Baseline: number analyzed (Participants) | 6 | 4 | 20 | 11
  Baseline | 46.838 (7.8986) | 43.118 (16.3701) | 37.071 (12.2914) | 39.512 (15.4212)
  Week 12: number analyzed (Participants) | 8 | 4 | 18 | 11
  Week 12 | 48.076 (12.5197) | 43.660 (13.9997) | 44.688 (10.2469) | 43.785 (13.2982)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 4 | 17 | 11
  Change from Baseline to Week 12 | 0.373 (6.3174) | 0.543 (4.0309) | 8.212 (11.1378) | 4.273 (10.7671)
Statistical Analysis 1: Comparison: Cohort 1 CFZ533 vs Cohort 1 Placebo; Test type: Superiority; p = 0.986, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-8.49 to 8.35]
Statistical Analysis 2: Comparison: Cohort 2 CFZ533 vs Cohort 2 Placebo; Test type: Superiority; p = 0.175, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 3.83, 95% CI 2-sided [-1.81 to 9.48]

7. Secondary Outcome: Change From Baseline in Multidimensional Fatigue Inventory (MFI)
Description: The MFI is a patient self-reported outcome measure (questionnaires) to assess fatigue covering the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Each dimension has a possible range from 4-20. The reported total score has a range from 20-100. A reduction from baseline in MFI indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo
Number analyzed (Participants) | 8 | 4 | 21 | 11
units on a scale
  Baseline: number analyzed (Participants) | 6 | 4 | 20 | 11
  Baseline | 54.1 (16.23) | 78.0 (17.80) | 70.0 (17.51) | 66.2 (17.59)
  Week 12: number analyzed (Participants) | 8 | 4 | 18 | 11
  Week 12 | 53.5 (13.96) | 69.8 (17.75) | 55.2 (16.65) | 63.3 (16.99)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 4 | 17 | 11
  Change from Baseline to Week 12 | -0.6 (8.12) | -8.3 (8.18) | -14.5 (18.09) | -2.9 (12.37)
Statistical Analysis 1: Comparison: Cohort 1 CFZ533 vs Cohort 1 Placebo; Test type: Superiority; p = 0.807, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.34, 95% CI 2-sided [-10.48 to 13.15]
Statistical Analysis 2: Comparison: Cohort 2 CFZ533 vs Cohort 2 Placebo; Test type: Superiority; p = 0.074, Repeated measures model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -9.83, 95% CI 2-sided [-20.66 to 1.01]

ADVERSE EVENTS:
Time Frame: Cohort 1 and 2: 255 days (30 days post study completion) Cohort 3: 171 days (30 days post study completion)
Arm/Group | Cohort 1 CFZ533 | Cohort 1 Placebo | Cohort 2 CFZ533 | Cohort 2 Placebo | Cohort 3 CFZ533 Arm 1 | Cohort 3 CFZ533 Arm 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/21 | 0/11 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/4 | 1/21 | 0/11 | 0/13 | 1/12
Other Adverse Events (participants affected / at risk) | 8/8 | 4/4 | 11/21 | 7/11 | 12/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 CFZ533 (N=8) | Cohort 1 Placebo (N=4) | Cohort 2 CFZ533 (N=21) | Cohort 2 Placebo (N=11) | Cohort 3 CFZ533 Arm 1 (N=13) | Cohort 3 CFZ533 Arm 2 (N=12)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 CFZ533 (N=8) | Cohort 1 Placebo (N=4) | Cohort 2 CFZ533 (N=21) | Cohort 2 Placebo (N=11) | Cohort 3 CFZ533 Arm 1 (N=13) | Cohort 3 CFZ533 Arm 2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 1
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nail bed infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 4
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 2 | 2 | 4 | 2
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 2
Urogenital infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal wall neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 1 | 2 | 4
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Endometrial disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT02291029/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT02291029/SAP_001.pdf